CLINICAL TRIAL: NCT00279604
Title: Targeted Interventions in Cannabis Abuse: Focus on Decision Making (INCA)
Brief Title: INCA - Intervention and Neuropsychology in Cannabis Abuse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01EB0432
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse

INTERVENTIONS:
Behavioral: 'Problem Profile Intervention' vs. WHO-Brief Intervention

SUMMARY:
INCA (Intervention and Neuropsychology of Cannabis Abuse) is a study combining two research goals. One is to study efficacy of a short intervention the 'Problem Profile Intervention', which utilizes individual feedback from a 'substance problem check-up'. Subjects will randomly receive the 'Problem Profile Intervention' or the WHO Brief Intervention, a brief intervention, which has been shown to be efficacious. Currently efficiency studies are under way. The WHO Brief Intervention has been translated into German by our group. In contrast to most other cannabis intervention studies the current study is focussed on cannabis abusers not so much cannabis-dependent subjects. A total of 160 subjects are to be recruited. Half of them will randomly receive either the Problem Profile Intervention or the WHO Brief Intervention (active control). A total of 25% of subjects from each group will be placed on a 3 months waiting list before receiving the intervention (inactive control). Intervention outcome will be assessed three months, six month and 12 months after the intervention. We hypothesize cannabis use to be reduced by 25% by the 'Problem Profile Intervention'. The second aim of the study is to study mechanism of substance abuse. Initial results from own studies and data from other groups point to executive cognitive functions as a subtle but important factor that can be compromised in cannabis users (Verdejo-Garcia et al., 2004; Garavan and Stout, 2005). Using an fMRI-study, we intend to examine a subgroup of our subjects on a specific aspect of executive functioning that has recently received major interest in drug research: Decision-making capability, or risk-taking behaviour, respectively (e.g. Ernst and Paulus, 2005).

ELIGIBILITY:
Inclusion Criteria:

* ASSIST-Score for cannabis consume ≥ 4 ≤ 26
* german mother tongue (or comparable level)

Exclusion Criteria:

* major current psychiatric disorder (e.g. psychosis)
* addiction to other illegal drugs or alcohol
* recent or current intravenous drug use
* CNS-affecting medication
* current psychotherapy, other treatment for substance use disorder

exclusion criteria for fMRI-part:

* left-handedness
* medication (birth control pill, thyroid gland hormones possible)
* internistic illnesses (hypertension, diabetes, diseases of lungs)
* metallic implants (cardiac pacemaker, ferromagnetic object implanted through surgical intervention or accident, large-area tattoos)
* history of serious trauma
* claustrophobia
* gestation

Ages: 16 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160
Dates: Start 2005-07; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Cannabis consumption,
motivational change

SECONDARY OUTCOMES:
ASSIST-Score

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Schuetz, MD MPH, Principal Investigator — University of Bonn, Department of Psychiatry
Locations (2):
- Germany (2):
  - Friedrich-Wilhelms-University, Department of Psychiatry, Bonn, North Rhine-Westphalia
  - University of Essen, Department of Psychiatry and Psychotherapy, Essen, North Rhine-Westphalia